CLINICAL TRIAL: NCT04770753
Title: A Phase 3, Double-Blind, Randomized, Placebo-Controlled, Multicenter Study Evaluating the Efficacy and Safety of Mitapivat in Subjects With Non-Transfusion-Dependent Alpha- or Beta-Thalassemia (ENERGIZE)
Brief Title: A Study Evaluating the Efficacy and Safety of Mitapivat in Participants With Non-Transfusion-Dependent Alpha- or Beta-Thalassemia (α- or β-NTDT)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG348-C-017; 2021-000211-23 (EudraCT Number)
Record Dates: First submitted 2021-02-18; First posted 2021-02-25 (Actual); Results first posted 2025-01-24 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Non-Transfusion-dependent Alpha-Thalassemia; Non-Transfusion-dependent Beta-Thalassemia
MeSH Terms: interventions — mitapivat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mitapivat (Experimental): Mitapivat 100 milligrams (mg), orally, twice daily (BID) for 24 weeks in double blind (DB) period and for up to 5 years in open label extension (OLE) period.
  Interventions: Drug: Mitapivat
- Placebo (Placebo Comparator): Placebo matching mitapivat, orally, BID for 24 weeks in double blind period followed by Mitapivat 100 mg, orally, BID for up to 5 years in open label extension period.
  Interventions: Drug: Placebo Matching Mitapivat; Drug: Mitapivat

INTERVENTIONS:
Drug: Placebo Matching Mitapivat — Tablets
  Arms: Placebo
Drug: Mitapivat — Tablets
  Other Names: AG-348; AG-348 sulfate hydrate; Mitapivat sulfate

SUMMARY:
The primary purpose of this study was to compare the effect of mitapivat versus placebo on hemolytic anemia in participants with alpha- or beta-non-transfusion dependent thalassemia (NTDT).

DETAILED DESCRIPTION:
The mitapivat group included 130 participants whereas the placebo group had 64 participants.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of thalassemia (β-thalassemia with or without α-globin gene mutations, hemoglobin E (HbE)/β-thalassemia, or α-thalassemia/hemoglobin H [HbH] disease) based on Hb electrophoresis, Hb high-performance liquid chromatography (HPLC)), and/or deoxyribonucleic acid (DNA) analysis;
* Hb concentration ≤10.0 grams per deciliter (g/dL) (100.0 grams per liter [g/L]), based on an average of at least 2 Hb concentration measurements (separated by ≥7 days) collected during the Screening Period;
* Non-transfusion-dependent, defined as ≤5 red blood cell (RBC) units during the 24-week period before randomization; and no RBC transfusions ≤8 weeks before providing informed consent and no RBC transfusions during the Screening Period;
* If taking hydroxyurea, the hydroxyurea dose must be stable for ≥16 weeks before randomization;
* Women of child-bearing potential (WOCBP) must be abstinent of sexual activities that may result in pregnancy as part of their usual lifestyle or agree to use 2 forms of contraception, one of which must be considered highly effective, from the time of providing informed consent, throughout the study, and for 28 days after the last dose of study drug. The second form of contraception can be an acceptable barrier method;
* Written informed consent before any study-related procedures are conducted and willing to comply with all study procedures for the duration of the study.

Exclusion Criteria:

* Pregnant, breastfeeding, or parturient
* Documented history of homozygous or heterozygous sickle hemoglobin (HbS) or hemoglobin C (HbC);
* Prior exposure to gene therapy or prior bone marrow or stem cell transplantation;
* Currently receiving treatment with luspatercept; the last dose must have been administered ≥18 weeks before randomization;
* Currently receiving treatment with hematopoietic stimulating agents; the last dose must have been administered ≥18 weeks before randomization;
* History of malignancy, (active or treated) ≤5 years before providing informed consent;
* History of active and/or uncontrolled cardiac or pulmonary disease ≤6 months before providing informed consent, except for nonmelanomatous skin cancer in situ, cervical carcinoma in situ, or breast carcinoma in situ;
* Hepatobiliary disorders;
* Estimated glomerular filtration rate <45 milliliters per minute (mL/min)/1.73 m^2 by Chronic Kidney Disease Epidemiology Collaboration creatinine equation;
* Nonfasting triglycerides >440 milligrams per deciliter (mg/dL) (5 millimoles per liter [mmol/L]);
* Active infection requiring systemic antimicrobial therapy at the time of providing informed consent;
* Positive test for hepatitis C virus antibody (HCVAb) with evidence of active HCV infection, or positive test for hepatitis B surface antigen (HBsAg);
* Positive test for human immunodeficiency virus (HIV)-1 antibody (Ab) or HIV-2 Ab;
* History of major surgery (including splenectomy) ≤16 weeks before providing informed consent and/or a major surgical procedure planned during the study;
* Current enrollment or past participation (≤12 weeks before administration of the first dose of study drug or a timeframe equivalent to 5 half-lives of the investigational study drug, whichever is longer) in any other clinical study involving an investigational treatment or device;
* Receiving strong CYP3A4/5 inhibitors that have not been stopped for ≥5 days or a timeframe equivalent to 5 half-lives (whichever is longer); or strong CYP3A4 inducers that have not been stopped for ≥4 weeks or a timeframe equivalent to 5 half-lives (whichever is longer), before randomization;
* Receiving anabolic steroids that have not been stopped for at least 4 weeks before randomization. Testosterone replacement therapy to treat hypogonadism is allowed. The testosterone dose and preparation must be stable for ≥10 weeks before randomization;
* Known allergy to mitapivat or its excipients (microcrystalline cellulose, croscarmellose sodium, sodium stearyl fumarate, mannitol, and magnesium stearate, Opadry® II Blue [hypromellose, titanium dioxide, lactose monohydrate, triacetin, and FD&C Blue #2]);
* Any medical, hematological, psychological, or behavioral condition(s) or prior or current therapy that, in the opinion of the Investigator, may confer an unacceptable risk to participating in the study and/or could confound the interpretation of the study data Also excluded are:

  * Participants who are institutionalized by regulatory or court order
  * Participants with any condition(s) that could create undue influence (including but not limited to incarceration, involuntary psychiatric confinement, and financial or familial affiliation with the Investigator or Sponsor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2028-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Chair — Agios Pharmaceuticals, Inc.
Locations (68):
- United States (6):
  - San Diego Hospital, UC San Diego Health, La Jolla, California
  - Stanford Medicine, Palo Alto, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Weill Cornell Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Penn Medicine - University of Pennsylvania Health System, Philadelphia, Pennsylvania
- Brazil (6):
  - Universidade de Caxias do Sul, Caxias do Sul
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto - USP, Ribeirão Preto
  - HEMORIO Instituto Nacional de Hematologia, Rio de Janeiro
  - Praxis Pesquisa Medica, Santo André
  - GSH Banco de Sangue de São Paulo, São Paulo
  - Instituto do Cancer do Estado de São Paulo, Hospital das Clínicas da Faculdade de Medicina da Universidad de São Paulo, São Paulo
- Bulgaria (2):
  - MHAT "Dr. Nikola Vasiliev" AD, Kyustendil
  - SHATHD Sofia, Sofia
- Toronto General Hospital, University Health Network, Toronto, Canada
- Rigshospitalet, Copenhagen, Denmark
- France (2):
  - CHU Hôpital Henri Mondor, Créteil
  - Hopital Edouard Herriot, CHU de Lyon, Lyon
- Greece (4):
  - Laiko General Hospital, Athens
  - Children's Hospital Agia Sophia, National and Kapodistrian University of Athens Medical School, Athens
  - University General Hospital of Patras, Rio
  - Ippokrateio General Hospital, Thessaloniki
- Italy (9):
  - Ospedale "A. Perrino" - Brindisi, Brindisi
  - Ospedale Pediatrico Microcitemico, Cagliari
  - Ospedale Sant'Anna, Ferrara
  - Ente Ospedaliero Ospedali Galliera, Genova
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - A.O.U Di Modena, Modena
  - A.O.R.N. "A. Cardarelli", Napoli
  - AOU L. Vanvitelli Universita degli Studi della Campania Luigi Vanvitelli, Napoli
  - A.O.U. San Luigi Gonzaga, Orbassano
- Chronic Care Center, Beirut, Lebanon
- Malaysia (8):
  - Hospital Sultanah Bahiyah, Alor Star
  - Hospital Ampang, Ampang
  - Hospital Sultanah Aminah Johor Bahru, Johor Bahru
  - Hospital Queen Elizabeth, Kota Kinabalu, Kota Kinabalu
  - Hospital Tunku Azizah, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Hospital Umum Sarawak, Kuching
  - Hospital Pulau Pinang, Pulau Pinang
- Netherlands (2):
  - Erasmus MC, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Saudi Arabia (2):
  - King Abdulaziz Hospital - Al Ahsa, Al Mubarraz
  - King Abdullah International Medical Research Center, Riyadh
- Spain (4):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen Arrixaca, Murcia
  - Hospital Universitario Virgen del Rocío, Seville
- China Medical University, Taiwan, Taichung, Taiwan
- Thailand (7):
  - Phramongkutklao Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Faculty of Medicine Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Srinagarind Hospital, Khon Kaen University, Khon Kaen
  - Naresuan University Hospital, Mueang Phitsanulok
  - King Chulalongkorn Memorial Hospital, Pathum Wan
- Turkey (Türkiye) (6):
  - Acibadem Adana Hospital, Adana
  - Akdeniz University Faculty of Medicine, Antalya
  - Çukurova University, Balcalı
  - Ege University Faculty of Medicine, Bornova
  - Istanbul University Faculty of Medicine, Fatih
  - Hacettepe University, Mersin
- United Arab Emirates (2):
  - Burjeel Medical City, Abu Dhabi
  - Thalassemia Centre Dubai, Dubai
- United Kingdom (4):
  - Cambridge University Hospitals NHS Foundation Trust - Addenbrookes Hospital, Cambridge, CAM
  - Manchester Royal Infirmary, Manchester University NHS Foundation Trust, Manchester, LAN
  - University College London, London
  - Imperial College Healthcare NHS Trust - Hammersmith Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taher AT, Al-Samkari H, Aydinok Y, Besser M, Boscoe AN, Dahlin JL, De Luna G, Estepp JH, Gheuens S, Gilroy KS, Glenthoj A, Sim Goh A, Iyer V, Kattamis A, Loggetto SR, Morris S, Musallam KM, Osman K, Ricchi P, Salido-Fierrez E, Sheth S, Tai F, Tevich H, Uhlig K, Urbstonaitis R, Viprakasit V, Cappellini MD, Kuo KHM; ENERGIZE investigators. Mitapivat in adults with non-transfusion-dependent alpha-thalassaemia or beta-thalassaemia (ENERGIZE): a phase 3, international, randomised, double-blind, placebo-controlled trial. Lancet. 2025 Jul 5;406(10498):33-42. doi: 10.1016/S0140-6736(25)00635-X. Epub 2025 Jun 19. PMID 40544857

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in study at study sites in the United States of America, Brazil, Bulgaria, Canada, Denmark, France, Greece, Italy, Lebanon, Malaysia, Netherlands, Saudi Arabia, Spain, Taiwan, Thailand, Turkey, United Arab Emirates and the United Kingdom. Results are reported for 24-week DB period until primary completion date. Analysis of data for OLE period is still ongoing with anticipated completion in December 2028. Results for OLE period will be reported by December 2029.
Pre-assignment Details: A total of 235 participants with a diagnosis of Non-Transfusion-Dependent Alpha- or Beta-Thalassemia (α- or β-NTDT) were screened. Of which, 194 were enrolled and 192 were treated in this study.
Groups:
- Mitapivat: Participants randomized to receive Mitapivat 100 milligrams (mg), orally, twice daily (BID) for 24 weeks in double blind period and for up to 5 years in open label extension period.
- Placebo: Participants randomized to receive placebo matching mitapivat, orally, BID for 24 weeks in double blind period followed by Mitapivat 100 mg, orally, BID for up to 5 years in open label extension period.
Period: Overall Study
Arm/Group | Mitapivat | Placebo
Started | 130 | 64
Treated | 129 | 63
Completed | 122 | 62
Not Completed | 8 | 2
Not completed — Randomized, never treated | 1 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Other un-specified | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mitapivat | Placebo | Total
Number analyzed (Participants) | 130 | 64 | 194
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (13.03) | 38.9 (12.99) | 41.2 (13.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 39 | 123
  Male | 46 | 25 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 6 | 17
  Not Hispanic or Latino | 118 | 58 | 176
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 73 | 36 | 109
  Asian | 52 | 24 | 76
  Black or African American | 1 | 1 | 2
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Multiracial | 1 | 0 | 1
  Unknown | 2 | 2 | 4
  Not reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Double-Blind Period: Percentage of Participants Who Achieved Hemoglobin (Hb) Response From Week 12 Through Week 24 Compared With Baseline
Description: Hb response is defined as ≥10 grams/ liter (g/L) (1.0 gram per deciliter) (g/dL) increase in average Hb concentration from Week 12 through Week 24 compared with baseline. Hb response was tested using the Mantel-Haenszel stratum weighted method adjusting for randomization stratification factors. Baseline is defined as the average of all assessments within 42 days before randomization for subjects randomized and not dosed or within 42 days before the start of study treatment for subjects randomized and dosed.
Time Frame: Double-Blind Period: Baseline up to Week 12 through Week 24
Population: FAS included all participants who were randomized.
Measure: Number; unit: Percentage of participants
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 130 | 64
Percentage of participants | 42.3 | 1.6
Statistical Analysis 1: Comparison: Mitapivat vs Placebo; The estimated adjusted difference in response rate, 95% CI, and p-value are based on Mantel-Haenszel stratum weighted method adjusting for the randomization stratification factors; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Percentage difference = 40.9, 95% CI 2-sided [32.0 to 49.8]

2. Secondary Outcome: Double-Blind Period: Change From Baseline in Average Functional Assessment of Chronic Illness Therapy (FACIT) -Fatigue Subscale Score From Week 12 Through Week 24
Description: The FACIT-Fatigue subscale includes a 13-item self-reported fatigue subscale, which assesses the severity and impact of fatigue (including the impact on daily activities and functioning).The FACIT-Fatigue subscale is scored on a 5-point Likert scale: 0 (not at all) to 4 (very much). The total FACIT-Fatigue subscale score ranges from 0 to 52, with a higher score indicating better health-related quality of life (HRQOL). Baseline is defined as the last assessment before randomization for subjects randomized and not dosed or the last assessment before start of study treatment for subjects randomized and dosed.
Time Frame: Double-Blind Period: Baseline, Week 12 through Week 24
Population: FAS included all participants who were randomized. Overall number of participants analyzed indicates number of participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 109 | 54
score on a scale | 4.85 (0.732) | 1.46 (0.955)
Statistical Analysis 1: Comparison: Mitapivat vs Placebo; The estimates, 95% CIs, and 2-sided p-value are based on an analysis of covariance (ANCOVA) model which includes average change from baseline in FACIT-Fatigue subscale score from Week 12 through Week 24 as the dependent variable, treatment group as the independent variable, and baseline and the randomization stratification factors as covariates; Test type: Superiority; p = 0.0026, ANCOVA; Difference in Lean Square (LS) Mean = 3.40, 95% CI 2-sided [1.21 to 5.59]

3. Secondary Outcome: Double-Blind Period: Change From Baseline in Average Hb Concentration From Week 12 Through Week 24
Description: Baseline is defined as the average of all assessments within 42 days before randomization for subjects randomized and not dosed or within 42 days before the start of study treatment for subjects randomized and dosed.
Time Frame: Double-Blind Period: Baseline, Week 12 through Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Gram per Liter (g/L)
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 123 | 61
Gram per Liter (g/L) | 8.57 (0.666) | -1.06 (0.867)
Statistical Analysis 1: Comparison: Mitapivat vs Placebo; The estimates, 95% CIs, and 2-sided p-value are based on an ANCOVA model which includes average change from baseline in Hb concentrations from Week 12 through Week 24 as the dependent variable, treatment group as the independent variable, and baseline Hb concentration and the randomization stratification factors as covariates; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LS Mean = 9.63, 95% CI 2-sided [7.80 to 11.46]

4. Secondary Outcome: Double-Blind Period: Percentage of Participants Who Achieved Hb 1.5+ Response From Week 12 Through Week 24 Compared With Baseline
Description: Hb 1.5+ response is defined as a ≥1.5 g/dL increase in average Hb concentration from Week 12 through Week 24 compared with baseline. Hb 1.5+ response will be summarized using the Mantel-Haenszel stratum weighted method adjusting for randomization stratification factors. Baseline is defined as the average of all assessments within 42 days before randomization for subjects randomized and not dosed or within 42 days before the start of study treatment for subjects randomized and dosed.
Time Frame: Double-Blind Period: Baseline up to Week 12 through Week 24
Population: FAS included all participants who were randomized.
Measure: Number; unit: Percentage of participants
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 130 | 64
Percentage of participants | 24.6 | 0

5. Secondary Outcome: Double-Blind Period: Change From Baseline in Indirect Bilirubin at Week 24
Description: as for outcome 3
Time Frame: Double-Blind Period: Baseline, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Micromole per Liter (umol/L)
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 116 | 54
Micromole per Liter (umol/L) | -10.65 (1.047) | -0.03 (1.403)

6. Secondary Outcome: Double-Blind Period: Change From Baseline in Lactate Dehydrogenase (LDH) at Week 24
Description: as for outcome 3
Time Frame: Double-Blind Period: Baseline, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units per Liter (U/L)
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 116 | 54
Units per Liter (U/L) | -30.07 (7.131) | -5.79 (9.440)

7. Secondary Outcome: Double-Blind Period: Change From Baseline in Haptoglobin at Week 24
Description: as for outcome 3
Time Frame: Double-Blind Period: Baseline, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Gram per Liter (g/L)
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 115 | 55
Gram per Liter (g/L) | -0.002 (0.0145) | 0.017 (0.0199)

8. Secondary Outcome: Double-Blind Period: Change From Baseline in Reticulocytes at Week 24
Description: as for outcome 3
Time Frame: Double-Blind Period: Baseline, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: 10^9 cells per liter (10^9 cells/L)
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 86 | 37
10^9 cells per liter (10^9 cells/L) | -32.11 (10.600) | -14.74 (14.932)

9. Secondary Outcome: Double-Blind Period: Change From Baseline in Erythropoietin at Week 24
Description: as for outcome 3
Time Frame: Double-Blind Period: Baseline, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: International units per Liter (IU/L)
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 103 | 47
International units per Liter (IU/L) | 19.21 (37.773) | 115.71 (49.413)

10. Secondary Outcome: Double-Blind Period: Percentage of Participants Who Achieved Patient Global Impression of Severity (PGIS)- Fatigue Response at Weeks 12, 16, 20, and 24
Description: PGIS-Fatigue measured participants' perception of their fatigue severity (7-day recall) on a 4-point scale ranging from '1=none' to '4=severe'. A participant was considered to have achieved the PGIS-Fatigue response at Weeks 12, 16, 20, or 24, if their baseline to postbaseline score met one of the following conditions: 'none' at baseline to 'none' postbaseline; 'mild' to 'mild' or 'none'; 'moderate' to 'mild' or 'none'; or 'severe' to 'moderate', 'mild', or 'none'.
Time Frame: Double-Blind Period: At Weeks 12, 16, 20, and 24
Population: FAS included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 130 | 64
percentage of participants
  At Week 12 | 65.4 | 46.9
  At Week 16 | 63.1 | 42.2
  At Week 20 | 61.5 | 48.4
  At Week 24 | 62.3 | 46.9

11. Secondary Outcome: Double-Blind Period: Percentage of Participants Who Achieved the Patient Global Impression of Change (PGIC)- Fatigue Response at Weeks 12, 16, 20, and 24
Description: The PGIC-Fatigue assesses change over time compared with baseline on a 5-point scale ranging from 0 to 4 where 0 indicates Much better and 4 as Much worse. A participant was considered to have achieved the PGIC-Fatigue response at Weeks 12, 16, 20, or 24 if their baseline PGIS and corresponding PGIC met one of the following conditions: if the PGIS at baseline was 'none' or 'mild' and PGIC at the visit was 'no change', 'a little better', or 'much better'; or if the PGIS at baseline was 'moderate' or 'severe' and PGIC at the visit was 'a little better' or 'much better'.
Time Frame: Double-Blind Period: At Weeks 12, 16, 20, and 24
Population: FAS included all participants who were randomized.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Participants randomized to receive placebo matching mitapivat, orally, BID for 24 weeks in double blind period followed by Mitapivat 100 mg, orally, BID for 5 up to years in open label extension period.
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 130 | 64
percentage of participants
  At Week 12 | 71.5 | 53.1
  At Week 16 | 71.5 | 50.0
  At Week 20 | 66.2 | 56.3
  At Week 24 | 66.2 | 53.1

12. Secondary Outcome: Double-Blind Period: Change From Baseline in the 6-minute Walk Test (6MWT) Distance at Week 24
Description: The 6MWT is a well-established performance outcome (PerfO) measure that is widely used to evaluate physical activity in terms of distance walked in patients with a variety of conditions. The test measures the distance an individual can walk on a hard, flat surface in 6 minutes.
Time Frame: Double-Blind Period: Baseline, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Meters
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 107 | 57
Meters | 30.48 (5.651) | 7.11 (7.346)

13. Secondary Outcome: Double-Blind Period: Change From Baseline in Serum Ferritin at Week 24
Description: Iron metabolism was assessed based on serum ferritin levels.
Time Frame: Double-Blind Period: Baseline, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Microgram/Liter (mcg/L)
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 116 | 56
Microgram/Liter (mcg/L) | -34.75 (32.710) | -32.48 (43.090)

14. Secondary Outcome: Double-Blind Period: Change From Baseline in Transferrin Saturation (TSAT) at Week 24
Description: Iron metabolism was assessed based on TSAT levels. Transferrin saturation is reported by dividing value of serum iron by total iron binding capacity.
Time Frame: Double-Blind Period: Baseline, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 72 | 40
Ratio | -0.029 (0.0212) | -0.047 (0.0262)

15. Secondary Outcome: Double-Blind Period: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, Related TEAEs and TEAEs With Severity Greater Than or Equal to Grade 3
Description: AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with the study drug. A serious adverse event (SAE) is any untoward medical occurrence that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs are AEs with an initial onset date during the on-treatment period or worsening from baseline and includes both serious & non-serious TEAEs. Severity of AEs was evaluated using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE; Version 4.03): grade 1: mild; grade 2: moderate; grade 3: severe or medically significant but not immediately life-threatening; grade 4: life threatening or disabling; grade 5: death related to AE.
Time Frame: Double-Blind Period: From the time of signing informed consent to Week 24
Population: Safety Analysis Set (SAS) includes all participants who had received at least 1 dose of study treatment. Participants were classified according to the treatment received. If a participant was randomized to placebo and received at least 1 dose of mitapivat in the Double-blind Period, then the participant was classified to the mitapivat arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 129 | 63
Participants
  Participants with TEAEs | 107 | 50
  Participants with Serious TEAEs | 8 | 0
  Participants with TEAEs related to study drug | 56 | 13
  Participants with any TEAE of Grade ≥ 3 | 18 | 2

16. Secondary Outcome: Double-Blind Period: Plasma Concentration of Mitapivat
Time Frame: Double-Blind Period: Pre-dose at Week 12; pre-dose, 0.5, 1, 3, 5, 7 hours post-dose at Week 20
Population: Pharmacokinetic (PK) Analysis Set included a subset of the safety analysis set including all subjects with at least 1 mitapivat plasma concentration measurement ≥LLQ (lower limit of quantification). Number analyzed signifies those participants who were evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Mitapivat
Number analyzed (Participants) | 124
nanograms per milliliter (ng/mL)
  Pre-dose at Week 12: number analyzed (Participants) | 100
  Pre-dose at Week 12 | 59.23 (51.081)
  Pre-dose at Week 20: number analyzed (Participants) | 118
  Pre-dose at Week 20 | 84.70 (138.852)
  30 Minutes Post-dose at Week 20: number analyzed (Participants) | 119
  30 Minutes Post-dose at Week 20 | 1209.00 (931.211)
  1 Hour Post-dose at Week 20: number analyzed (Participants) | 118
  1 Hour Post-dose at Week 20 | 1386.35 (712.996)
  3 Hour Post-dose at Week 20: number analyzed (Participants) | 120
  3 Hour Post-dose at Week 20 | 740.26 (357.660)
  5 Hour Post-dose at Week 20: number analyzed (Participants) | 117
  5 Hour Post-dose at Week 20 | 359.42 (269.758)
  7 Hour Post-dose at Week 20: number analyzed (Participants) | 114
  7 Hour Post-dose at Week 20 | 206.82 (185.657)

17. Secondary Outcome: Double-Blind Period: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Measurable Concentration (AUC0-last) of Mitapivat
Description: Area under the concentration-time curve from time zero to Tlast on dosing day, calculated using the linear-log trapezoidal rule.
Time Frame: Double-Blind Period: Pre-dose, 0.5, 1, 3, 5, 7 hours post-dose at Week 20
Population: Pharmacokinetic (PK) Analysis Set included a subset of the safety analysis set including all subjects with at least 1 mitapivat plasma concentration measurement ≥LLQ. Overall number of participants analyzed indicates number of participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter (h*ng/mL)
Arm/Group | Mitapivat
Number analyzed (Participants) | 114
Hours*nanogram per milliliter (h*ng/mL) | 4262.57 (31.4)

18. Secondary Outcome: Double-Blind Period: Time of Last Quantifiable Concentration (Tlast) of Mitapivat
Time Frame: Double-Blind Period: Pre-dose, 0.5, 1, 3, 5, 7 hours post-dose at Week 20
Population: as for outcome 17
Measure: Median (Full Range); unit: hours
Arm/Group | Mitapivat
Number analyzed (Participants) | 114
hours | 6.825 [6.50 to 7.42]

19. Secondary Outcome: Double-Blind Period: Maximum Observed Plasma Concentration (Cmax) of Mitapivat
Time Frame: Double-Blind Period: Pre-dose, 0.5, 1, 3, 5, 7 hours post-dose at Week 20
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Mitapivat
Number analyzed (Participants) | 121
ng/mL | 1565.69 (42.4)

20. Secondary Outcome: Double-Blind Period: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Mitapivat
Time Frame: Double-Blind Period: Pre-dose, 0.5, 1, 3, 5, 7 hours post-dose at Week 20
Population: as for outcome 17
Measure: Median (Full Range); unit: Hours
Arm/Group | Mitapivat
Number analyzed (Participants) | 121
Hours | 1.000 [0.20 to 5.00]

21. Secondary Outcome: Double-Blind Period: Last Quantifiable Plasma Concentration (Clast) of Mitapivat
Time Frame: Double-Blind Period: Pre-dose, 0.5, 1, 3, 5, 7 hours post-dose at Week 20
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Mitapivat
Number analyzed (Participants) | 121
ng/mL | 166.93 (80.1)

22. Secondary Outcome: Double-Blind Period: Blood Concentration of Adenosine Triphosphate (ATP)
Time Frame: Double-Blind Period: Pre-dose at Day 1; pre-dose at Week 12; pre-dose, 0.5, 1, 3, 5, 7 hours post-dose at Week 20
Population: Pharmacodynamic (PD) Analysis Set is a subset of the safety analysis set including all participants with at least 1 blood 2,3-DPG or ATP concentration measurement ≥ LLQ. Number analyzed signifies those participants who were evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: microgram/milliliter (mcg/mL)
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 122 | 59
microgram/milliliter (mcg/mL)
  At Pre-dose at Day 1: number analyzed (Participants) | 93 | 44
  At Pre-dose at Day 1 | 180.87 (29.577) | 184.91 (31.299)
  Pre-dose at Week 12: number analyzed (Participants) | 91 | 47
  Pre-dose at Week 12 | 242.07 (45.782) | 176.81 (33.657)
  Pre-dose at Week 20: number analyzed (Participants) | 105 | 51
  Pre-dose at Week 20 | 235.79 (46.099) | 168.10 (29.962)
  30 Minutes Post-dose at Week 20: number analyzed (Participants) | 105 | 45
  30 Minutes Post-dose at Week 20 | 417.87 (102.853) | 457.78 (89.932)
  1 Hour Post-dose at Week 20: number analyzed (Participants) | 104 | 48
  1 Hour Post-dose at Week 20 | 417.83 (105.752) | 457.71 (104.431)
  3 Hour Post-dose at Week 20: number analyzed (Participants) | 106 | 49
  3 Hour Post-dose at Week 20 | 409.73 (96.379) | 454.39 (107.966)
  5 Hour Post-dose at Week 20: number analyzed (Participants) | 101 | 49
  5 Hour Post-dose at Week 20 | 412.72 (94.150) | 464.24 (97.007)
  7 Hour Post-dose at Week 20: number analyzed (Participants) | 102 | 49
  7 Hour Post-dose at Week 20 | 404.43 (97.586) | 471.10 (113.165)

23. Secondary Outcome: Double-Blind Period: Blood Concentration of 2,3 - Diphosphoglycerate (2,3-DPG)
Time Frame: Double-Blind Period: Pre-dose at Day 1; pre-dose at Week 12; pre-dose, 0.5, 1, 3, 5, 7 hours post-dose at Week 20
Population: Pharmacodynamic (PD) Analysis Set is a subset of the safety analysis set including all participants with at least 1 blood 2,3-DPG or ATP concentration measurement ≥LLQ. Number analyzed signifies those participants who were evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 122 | 59
mcg/mL
  Pre-dose at Day 1: number analyzed (Participants) | 93 | 44
  Pre-dose at Day 1 | 526.40 (125.196) | 506.14 (108.033)
  Pre-dose at Week 12: number analyzed (Participants) | 91 | 47
  Pre-dose at Week 12 | 434.90 (97.901) | 497.68 (112.055)
  Pre-dose at Week 20: number analyzed (Participants) | 105 | 50
  Pre-dose at Week 20 | 426.30 (107.173) | 468.22 (99.783)
  30 Minutes Post-dose at Week 20: number analyzed (Participants) | 105 | 45
  30 Minutes Post-dose at Week 20 | 417.87 (102.853) | 457.78 (89.932)
  1 Hour Post-dose at Week 20: number analyzed (Participants) | 104 | 48
  1 Hour Post-dose at Week 20 | 417.83 (105.752) | 457.71 (104.431)
  3 Hour Post-dose at Week 20: number analyzed (Participants) | 106 | 49
  3 Hour Post-dose at Week 20 | 409.73 (96.379) | 454.39 (107.966)
  5 Hour Post-dose at Week 20: number analyzed (Participants) | 101 | 49
  5 Hour Post-dose at Week 20 | 412.72 (94.150) | 464.24 (97.007)
  7 Hour Post-dose at Week 20: number analyzed (Participants) | 102 | 49
  7 Hour Post-dose at Week 20 | 404.43 (97.586) | 471.10 (113.165)

24. Secondary Outcome: Open-Label Extension Period: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, Related TEAEs and TEAEs With Severity of Greater Than or Equal to Grade 3
Description: AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with the study drug. A serious adverse event (SAE) is any untoward medical occurrence that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs are AEs with an initial onset date during the on-treatment period or worsening from baseline and includes both serious & non-serious TEAEs. Severity of abnormalities was evaluated using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE; Version 4.03): grade 1: mild; grade 2: moderate; grade 3: severe or medically significant but not immediately life-threatening; grade 4: life threatening or disabling; grade 5: death related to AE.
Time Frame: Open-Label Extension Period: From week 24 up to end of study (approximately 5 years)
Reporting Status: Not Posted, anticipated posting 2029-12

ADVERSE EVENTS:
Time Frame: Double-blind period: From the time of signing informed consent to Week 24
Description: Adverse events: Safety analysis set was used. Participants classified according to treatment received. If participant was randomized to placebo & received at least 1 dose of mitapivat in Double-blind Period, then participant was classified to mitapivat arm. All-Cause Mortality: FAS was used. Safety data are presented for Double-blind Period only. The OLE period is ongoing with anticipated completion in December 2028. Results for OLE will be reported separately by December 2029.
Arm/Group | Mitapivat | Placebo
All-Cause Mortality (participants affected / at risk) | 0/130 | 0/64
Serious Adverse Events (participants affected / at risk) | 8/129 | 0/63
Other Adverse Events (participants affected / at risk) | 80/129 | 33/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mitapivat (N=129) | Placebo (N=63)
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Craniofacial fracture (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Superficial vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mitapivat (N=129) | Placebo (N=63)
Upper respiratory tract infection (Infections and infestations) | 13 | 4
COVID-19 (Infections and infestations) | 8 | 5
Influenza (Infections and infestations) | 5 | 6
Nausea (Gastrointestinal disorders) | 15 | 5
Diarrhoea (Gastrointestinal disorders) | 11 | 6
Initial insomnia (Psychiatric disorders) | 18 | 3
Middle insomnia (Psychiatric disorders) | 8 | 1
Insomnia (Psychiatric disorders) | 7 | 1
Headache (Nervous system disorders) | 29 | 6
Fatigue (General disorders) | 12 | 4
Pyrexia (General disorders) | 4 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2024-08-05): https://cdn.clinicaltrials.gov/large-docs/53/NCT04770753/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-14): https://cdn.clinicaltrials.gov/large-docs/53/NCT04770753/SAP_001.pdf